CLINICAL TRIAL: NCT06691555
Title: The Long-term Safety and Efficacy of a Modified Suprachoroidal Silicone Tube (SST) Shunt in Patients with Primary Open-angle Glaucoma (POAG) and Pseudo-exfoliative Glaucoma (PXG) Over an Extended Follow-up Period
Brief Title: Long-term Safety and Efficacy of a Modified Suprachoroidal Silicone Tube (SST) Shunt
Status: Recruiting | Type: Observational
Sponsor: Davinci LTD (Other)
Responsible Party: Sponsor
Other Study IDs: SCS_L_002
Record Dates: First submitted 2024-11-09; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Glaucoma; Open Angle Glaucoma (OAG); POAG; Ocular Hypertension; Exfoliation Syndrome; Choroidal Effusions
Keywords: MIGS; Suprachoroidal Space; Glaucoma; Open-Angle Glaucoma; Suprachoroidal Silicone Tube; Suprachoroidal Shunt; Glaucoma Shunt
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Ocular Hypertension; Exfoliation Syndrome; Choroidal Effusions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group 1 that includes Primary Open-Angle Glaucoma and Pseudoexfoliative Glaucoma Patients: This cohort includes patients diagnosed with primary open-angle glaucoma (POAG) and pseudoexfoliative glaucoma (PXG) who have undergone suprachoroidal silicone tube (SST) shunt implantation. The study focuses on assessing the long-term safety and efficacy of the SST shunt, monitoring intraocular pressure (IOP) control, endothelial cell count (ECC) changes, and any adverse events over an extended follow-up period. This observational cohort includes patients aged 41-88 years, treated with the SST shunt either alone or in combination with cataract surgery, and meeting the inclusion criteria from a prior retrospective study.
  Interventions: Device: Suprachoroidal silicone tube (SST) shunt

INTERVENTIONS:
Device: Suprachoroidal silicone tube (SST) shunt — This intervention involves implanting a modified suprachoroidal silicone tube (SST) shunt, derived from the Aurolab Aqueous Drainage Device (AADI), to lower intraocular pressure in patients with primary open-angle and pseudoexfoliative glaucoma. The SST shunt, measuring 13.0-15.0 mm with a 0.3 mm inner and 0.6 mm outer diameter, is designed to reach the posterior suprachoroidal space. Six slits near the distal end aid aqueous outflow. Implantation involves creating a scleral flap, accessing the SCS, and placing the distal end in the SCS and proximal end in the anterior chamber (AC). The shunt is secured with sutures, and viscoelastic is injected into the AC to prevent hypotony. No antimetabolites or cautery are used.

SUMMARY:
The goal of this observational study is to evaluate the long-term safety and efficacy of a modified suprachoroidal silicone tube (SST) shunt in treating patients with primary open-angle glaucoma (POAG) and pseudo-exfoliative glaucoma (PXG).

The main questions it aims to answer are:

Does the SST shunt maintain intraocular pressure (IOP) reduction over an extended follow-up period? What is the effect of the SST shunt on endothelial cell count (ECC) and overall corneal health?

Participants will:

Undergo intraocular pressure (IOP) measurements Have their endothelial cell count (ECC) evaluated Complete assessments of best corrected visual acuity (BCVA) Be assessed for C/D ratio Be monitored for adverse events or shunt-related complications over time

DETAILED DESCRIPTION:
This observational study serves as an extension to a prior retrospective cross-sectional trial that initially investigated the clinical outcomes of suprachoroidal silicone tube (SST) shunt implantation in patients diagnosed with primary open-angle glaucoma (POAG) and pseudoexfoliative glaucoma (PXG). In the initial study, participants underwent the SST shunt procedure and were followed for an average period of 19 months post-surgery. This initial study focused on assessing intraocular pressure (IOP) reduction and the initial safety profile of the SST device. However, as the device's long-term impact on ocular health, particularly the corneal endothelium, was not fully understood, this follow-up observational study was designed and implemented approximately 1 year after the last FU data collection was completed.

The SST shunt device is a relatively novel intervention positioned between minimally invasive glaucoma surgeries (MIGS) and traditional tube shunt surgeries. By facilitating aqueous humor drainage from the anterior chamber to the suprachoroidal space, the SST shunt provides a unique pathway for IOP reduction. Given the risks associated with corneal endothelial health in glaucoma patients, especially following invasive procedures, understanding the long-term impact of the SST shunt on endothelial cell counts (ECC) is essential.

Study Objectives:

The primary objective of this observational study is to evaluate the long-term safety and efficacy of the SST shunt in reducing IOP and preserving endothelial cell health. This involves:

Tracking changes in ECC attributable solely to the SST shunt, as the study design excluded additional interventions to isolate the device's effect.

Assessing the device's ability to maintain effective IOP control over an extended period.

Documenting any adverse events, including device migration, extrusion, and other complications, to understand the SST shunt's overall impact on ocular health.

Study Population:

The study is going to re-evaluate approximately 66 eyes, who had previously undergone SST shunt implantation, either as a standalone procedure or in combination with cataract surgery. These evaluations are going to be conducted within the period between 8 Nov/2024 and 30 Nov/2024.Participants in this observational study met the original inclusion criteria set forth in the retrospective trial. This included a cohort of Caucasian patients aged 41 to 88 years (mean age: 69), with a gender distribution of 40 men and 26 women. All patients were untreated with glaucoma surgeries or laser therapies prior to the SST implantation, providing a clean baseline for evaluating the SST device's isolated effects.

Study Design:

This study is observational and non-interventional, meaning it involved no additional treatments or manipulations beyond the baseline SST shunt implantation. This approach allowed for a naturalistic assessment of ECC and other clinical parameters over time. By not introducing any new variables, the study design aimed to observe and measure outcomes that could be directly attributed to the SST shunt. This design offers valuable insights into the natural progression of endothelial cell health and IOP management in patients who have undergone SST implantation without the influence of confounding factors.

Clinical Assessments and Follow-Up Procedures With an average 31 months (std. dev: 8 monts) follow-up, participants underwent assessments to monitor IOP, visual acuity, ECC, C/D ratio and any shunt-related adverse events.

Outcome Measures:

Primary Outcomes:

Endothelial Cell Loss: Tracked to assess corneal integrity. IOP Control: Success was defined as ≥20% reduction in IOP, with "complete success" for IOP control without medications, "qualified success" with medications, and "failure" for <20% IOP reduction or IOP >21 mmHg.

Secondary Outcomes:

Hypotony: Defined as IOP <5 mmHg, categorized as transient or permanent. Device Migration/Extrusion: Monitored to assess mechanical stability. Other Adverse Events: Any device-related complications documented for safety analysis.

ELIGIBILITY:
Inclusion Criteria:

* Previously were treated with Suprachoroidal silicone tube shunt
* Willing and able to participate in this cross sectional observational follow up
* Participant capable of giving informed consent

Exclusion Criteria:

* Condition that could impact the ability of the participant to attend a follow-up visit as per the discretion of the investigator

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is going to re-evaluate approximately 66 eyes, who had previously undergone SST shunt implantation, either as a standalone procedure or in combination with cataract surgery. These evaluations are going to be conducted within the period between 8 Nov/2024 and 30 Nov/2024.Participants in this observational study met the original inclusion criteria set forth in the retrospective trial. This included a cohort of Caucasian patients aged 41 to 88 years (mean age: 69), with a gender distribution of 40 men and 26 women. All patients were untreated with glaucoma surgeries or laser therapies prior to the SST implantation, providing a clean baseline for evaluating the SST device's isolated effects.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Endothelial Cell Loss | From enrollment to the end of long term observational FU (average duration is 31 months with 8 months std. dev)
IOP Control: Success was defined as ≥20% reduction in IOP, with "complete success" for IOP control without medications, "qualified success" with medications, and "failure" for <20% IOP reduction or IOP >21 mmHg. | From enrollment to the end of long term observational FU (average duration is 31 months with 8 months std. dev)

SECONDARY OUTCOMES:
Hypotony, defined as intraocular pressure (IOP) < 5 mmHg, categorized as either transient or permanent. | From enrollment to the end of long term observational FU (average duration is 31 months with 8 months std. dev)
Device migration or extrusion, monitored to assess mechanical stability of the implant. | From enrollment to the end of long term observational FU (average duration is 31 months with 8 months std. dev)
Adverse Events/Severe Adverse Events: Device-related or non-device-related | From enrollment to the end of long term observational FU (average duration is 31 months with 8 months std. dev)

CONTACTS AND LOCATIONS:
Locations (1):
- Davinci Eye Center, LTD, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: No